CLINICAL TRIAL: NCT05577793
Title: Effect of Therapeutic Touch and Mother's Voice on Pain and Comfort Level During Nasal CPAP Application in Turkey: A Randomized Controlled Study
Brief Title: Effect of Therapeutic Touch and Mother's Voice on Pain and Comfort Level During Nasal CPAP Application
Acronym: CPAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ayşe Belpınar (Other)
Responsible Party: Sponsor-Investigator, Ayşe Belpınar, Lecturer, Bozok University
Organization: Bozok University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ABelpinar
Record Dates: First submitted 2022-09-23; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Preterm Infants; Nasal Continuous Positive Airway Pressure; Pain Management
Keywords: Nasal continuous positive airway pressure (NCPAP); Therapeutic Touch; Mother's Voice; Pain; Comfort
MeSH Terms: conditions — Agnosia; Pain | interventions — Therapeutic Touch; Control Groups

STUDY DESIGN:
Intervention Model Description: This study used a randomized controlled trial. A parallel trial design was used describing three different experimental groups (Therapeutic Touch, Mother's Voice, and Therapeutic Touch+Mother's Voice) and a control group.
Who Masked: Participant
Masking Description: Because of the nature of the intervention, double-blinding was not possible in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mother's Voice (Experimental): The mothers were asked to sing lullabies, and their voices were recorded in a quiet environment. Which lullaby they would sing was left to the mothers' discretion, and the audio recording process took an average of 2-3 minutes. The voice recordings taken were applied for a total of 15 minutes before, during and after the nasal CPAP application.The NIPS and PICS scores were evaluated and recorded before, during and after the application.
  Interventions: Other: Therapeutic Touch; Other: Mother's Voice +Therapeutic Touch; Other: Control
- Therapeutic Touch (Experimental): Therapeutic touch was started 5 minutes before nasal prongs were placed, and was applied for 5 minutes during the application, and continued for another 5 minutes after the nasal prongs were placed. The method was applied for a total of 15 minutes as 5 minutes of hand resting, 5 minutes of gentle caressing and 5 more minutes of hand resting.The NIPS and PICS scores were evaluated and recorded before, during and after the application.
  Interventions: Other: Mother's Voice; Other: Mother's Voice +Therapeutic Touch; Other: Control
- Mother's Voice+Therapeutic Touch (Experimental): Both applications were applied together for 15 minutes.The NIPS and PICS scores were evaluated and recorded before, during and after the application.
  Interventions: Other: Mother's Voice; Other: Therapeutic Touch; Other: Control
- Control (No Intervention): The premature babies in the control group did not receive any intervention other than the hospital procedure.The NIPS and PICS scores were evaluated and recorded before, during and after the application.

INTERVENTIONS:
Other: Mother's Voice — The audio recording was made to listen to the baby for 15 minutes during the nasal CPAP application. The NIPS and PICS scores were evaluated and recorded before, during and after the application.
  Other Names: Mother's Voice Group
  Arms: Mother's Voice+Therapeutic Touch; Therapeutic Touch
Other: Therapeutic Touch — Therapeutic touch was started 5 minutes before nasal prongs were placed, and was applied for 5 minutes during the application, and continued for another 5 minutes after the nasal prongs were placed. The method was applied for a total of 15 minutes as 5 minutes of hand resting, 5 minutes of gentle caressing and 5 more minutes of hand resting.The NIPS and PICS scores were evaluated and recorded before, during and after the application.
  Other Names: Therapeutic Touch Group
  Arms: Mother's Voice; Mother's Voice+Therapeutic Touch
Other: Mother's Voice +Therapeutic Touch — Both applications were applied together for 15 minutes.The NIPS and PICS scores were evaluated and recorded before, during and after the application.
  Other Names: Mother's Voice +Therapeutic Touch Group
  Arms: Mother's Voice; Therapeutic Touch
Other: Control — The premature babies in the control group did not receive any intervention other than the hospital procedure.The NIPS and PICS scores were evaluated and recorded before, during and after the application.
  Other Names: Control Group
  Arms: Mother's Voice; Mother's Voice+Therapeutic Touch; Therapeutic Touch

SUMMARY:
Aim: This study was conducted to evaluate the effects of Therapeutic Touch and Mother's Voice on pain and comfort levels of preterm infants during nasal CPAP application.

DETAILED DESCRIPTION:
Aim: This study was conducted to evaluate the effects of Therapeutic Touch and Mother's Voice on pain and comfort levels of preterm infants during nasal CPAP application.

Design and Method: The study, which used a randomized controlled trial, included 124 preterm neonatal infants a gestational age of 28- 37 weeks and received nasal CPAP. The infants were treated with Mother's Voice, Therapeutic Touch, and Mother's Voice+ Therapeutic Touch. The Neonatal Infant Pain Scale (NIPS) and Premature Infant Comfort Scale (PICS) scores of the infants were measured before, during and after the nasal CPAP application.

ELIGIBILITY:
Inclusion Criteria:

* being checked in at Neonatal Intensive Care Unit
* being in the gestational ages of 28 to 37 weeks
* having nasal CPAP

Exclusion Criteria:

* having neurological disorders
* having comorbidity
* receiving sedation or analgesics
* having congenital anomaly
* receiving extra invasive procedures or surgical intervention
* being diagnosed with hearing loss

Ages: 28 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 124 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2020-08-14 (Actual)

PRIMARY OUTCOMES:
Neonatal Infant Pain Scale (NIPS) | 15 minutes
  Neonatal Infant Pain Scale (NIPS) was developed by Lawrence et. al. in 1993 in order to assess intervention-related pain in term and preterm babies (Lawrence et al., 1993). The Turkish validity and reliability of the study was conducted in 1999 by Akdovan (Akdovan, 1999). NIPS has six sections on facial expression, crying, respiration state, movements of extremity, and being awake. All behavioral responses except for crying were given two separate scores (0-1 score). Three separate scores were assigned (0-1-2) to crying. The total scores were between 0-7. A high score showed that pain was more intense (Yilmaz & Arikan, 2011). The Cronbach's a coefficients before, during, and after the intervention were found to be 0.95, 0.87, and 0.88, respectively, by Lawrence et al. (Lawrence et al., 1993).The Neonatal Infant Pain Scale (NIPS) score was evaluated and recorded before, during and 15 minutes after the application.
Premature Infant Comfort Scale (PICS) | 15 minutes
  Premature Infant Comfort Scale (PICS) which was developed by Ambuel et. al. (Ambuel et al., 1992) in order to the measure pain and stress levels of 0-18-month-old children, was later adapted to 28-37-week-old premature infants by Monique et. al. in 2007 (Caljouw et al., 2007) The Premature Infant Comfort Scale assesses 7 parameters such as Awareness, Tranquility/Agitation, Respiration State (only supported by mechanical ventilation) or Crying (it was not assessed because it was scored only in children with spontaneous respiration), Physical Movement, Muscular Tonus, Facial Expressions and Average Cardiac Beat. The scale is 5-point Likert type. As the scale score increases, the comfort level decreases. The scores are between 35 and 7. Comfort decreases as it approaches 35 points, and increases as it approaches 7 points. (Küçük Alemdar & Güdücü Tüfekci, 2015).Premature Infant Comfort Scale (PICS) score was evaluated and recorded before, during and 15 minutes after the application.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Belpınar, Msc, Principal Investigator — Bozok University; Emriye Hilal Yayan, Phd, Principal Investigator — Inonu University
Locations (1):
- Cengiz Gökçek Gynecology, Obstetrics and Pediatrics Hospital, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No